CLINICAL TRIAL: NCT04681794
Title: Mayo Posture Positivity Power Program (MayoP4) for Active and Aging Individuals in Communities
Brief Title: Mayo Posture Positivity Power Program for Active and Aging Individuals in Communities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Takashi Nagai, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20-001520
Record Dates: First submitted 2020-10-21; First posted 2020-12-23 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Healthy Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MayoP4 Group (Experimental): MayoP4 is a 15-minute warmup with 4 different components of exercise: balance, posture, hopping/jumping, and movement-based mindfulness.
  Interventions: Other: exercise-based intervention
- Control Group (No Intervention): No intervention

INTERVENTIONS:
Other: exercise-based intervention — MayoP4 is a 15-minute warmup with 4 different components of exercise: balance, posture, jumping/hopping, and movement-based mindfulness.
  Other Names: MayoP4
  Arms: MayoP4 Group

SUMMARY:
The research is designed to answer effectiveness of community-based multimodal intervention programs on physical, mental, cognitive, social, and environmental in active and aging individuals.

DETAILED DESCRIPTION:
Despite that musculoskeletal diseases/conditions are the leading cause of disability and frailty/mortality in aging individuals, the musculoskeletal health is given little consideration. Exercise is essential and effective publicly-available medicine for management/prevention of obesity, lack of physical activity, chronic disease, frailty, and mental stress/anxiety/depression without any side-effects from drug use/abuse.

More recently, multimodal interventions with physical, postural, mindfulness, and power exercises have shown to be effective improving both physical and mental health. To expand the recent trend in multimodal intervention, the current proposal will examine effects of community-based multimodal intervention on physical, psychological, cognitive, social, and environmental characteristics in aging individuals. Simultaneously, a cross-sectional study will establish normative values and inter-relationships.

One simple (15 minutes a day /2-3 times a week) yet comprehensive multimodal (balance, posture/thoracic spine, hopping, and mindfulness) intervention could provide a practical solution for aging individuals. Such a program could be implemented individually or by community staff, which would allow for a large-scale community implementation.

Therefore, the overall objective of the project is to explore effects of a community-based, simple, multimodal intervention program (MayoP4) for aging individuals. A small group intervention with friends and club/family members will help peer-to-peer support/team spirit and improve positive engagement.

The secondary objective of this project is to establish normative values and examine interrelations among various frailty/mortality risk factors. In addition to physical activity, musculoskeletal, balance/posture, and psychological/wellness factors, there are many additional elements associated with frailty/mortality risk. These include, but are not limited to, positive thinking/behavior (optimism), sufficient sleep, and cognitive/social/environmental considerations. Physical frailty plays an important role and positively influences all other domains; however, this relationship among aging individuals in our communities remains to be established.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be physically capable (defined as easy to moderate physical activities daily at least 60 minutes).
* Participants also must have a normal (18.5-24.9kg/m2) or overweight BMI (25-29.9kg/m2).
* Participants must be able to speak, listen, read, and understand sentences written in English.

Exclusion Criteria:

* Participants who display more than two risk factors for coronary artery disease
* Participants who have a history of falls, osteoporosis, osteoarthritis, or orthopedic or neurological conditions (i.e., stroke)
* Participants who take medications that cause dizziness or slow movement
* Participants who smoke
* Participants who have a body mass to height squared ratio greater than 30kg/m2 or less than 18.4kg/m2, blood pressure greater than 140/90 mmHg, or a history of heart conditions.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 59 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline demographic information at 12 weeks | baseline, 12 weeks
  * Age (continuous),
  * Race (White, Black, Asian, Pacific Islander, Hispanic/Latino, American Indian)
  * Marital Status (married, divorced/separated/single, widowed)
  * Education (less than High School, High School, College, Graduate School)
  * Height
  * Weight
  * Smoking (never, former, current)
  * Alcohol (intake from wine, beer, and liquor - none, 1-14g/day, >15g/day.)
  * For Women Only: Women health questions will be asked for past/present conditions (pregnancy, hormonal treatment, menopause, supplements, medications, etc.)
Change from baseline frailty index information at 12 weeks, 1 | baseline, 12 weeks
  • Comprehensive Frailty Assessment Instrument Plus: Assessment of frailty in physical, psychological, social, cognitive, and environmental domains
Change from baseline Knee/Osteoarthritis Self-Reported Questionnaires at 12 weeks, 1 | baseline, 12 weeks
  • International Knee Documentation Committee Subjective Knee Evaluation
Changes from baseline psychological assessment at 12 weeks, 1 | baseline, 12 weeks
  • Perceived Stress Scale: A 14-item self-report tool that provides a global measure of perceived stress
Changes from baseline overall health surveys / physical frailty test at 12 weeks, 1 | baseline, 12 weeks
  • Medical Outcomes Study 36-Item Short-Form Health Survey: A common medical questionnaire for general health and wellbeing
Changes from baseline hand-Grip Strength at 12 weeks | baseline, 12 weeks
  A standard handgrip isometric strength test performed using a Jamar Hydraulic Hand Dynamometer.
Changes from baseline walking speed at 12 weeks | baseline, 12 weeks
  you will be asked to walk as fast as you can for 4-meter (12 feet) three times. 4-meter distance will be marked with a tape.
Changes from baseline knee strength at 12 weeks | baseline, 12 weeks
  A custom-built knee strength measuring device will examine your quadriceps muscles (front muscles of the thigh) and hamstrings muscles (back muscles of the thigh).
Changes from baseline knee muscular steadiness at 12 weeks | baseline, 12 weeks
  • Force steadiness test will assess individual's ability to hold their muscular force for 10 seconds steady.
Changes from baseline balance at 12 weeks | baseline, 12 weeks
  Standing balance with eyes-open and eyes-closed will be tested.
Changes from baseline posture at 12 weeks | baseline, 12 weeks
  standard 2D camera will be used to assess standing posture and overhead squatting posture.
Changes from baseline heel bone ultrasound scan at 12 weeks | baseline, 12 weeks
  Quantitative ultrasound is accurate, inexpensive, and portable alternative to DXA bone mineral density. This device will measure the speed of sound and the frequency-dependent attenuation of the sound waves to calculate the stiffness index which is equivalent to bone mineral density.
Changes from baseline ultrasound-based bilateral anterior thigh thickness at 12 weeks | baseline, 12 weeks
  A diagnostic musculoskeletal ultrasound will be used to measure your thigh muscle size.
Changes from baseline frailty index at 12 weeks, 2 | baseline, 12 weeks
  • A multi-domain frailty assessment
Changes from baseline knee/osteoarthritis self-reported questionnaires at 12 weeks, 2 | baseline, 12 weeks
  • Knee Osteoarthritis Outcome Score
Changes from baseline knee/osteoarthritis self-reported questionnaires at 12 weeks, 3 | baseline, 12 weeks
  • Knee Outcome Survey-Activities of Daily Living
Changes from baseline knee/osteoarthritis self-reported questionnaires at 12 weeks, 4 | baseline, 12 weeks
  • Global Rating score
Changes from baseline psychological assessment at 12 weeks, 2 | baseline, 12 weeks
  • Generalized Anxiety Disorder 7-item: A 7-item questionnaire which asks how often, during the last 2 weeks, the participant was bothered by anxiety-related symptoms
Changes from baseline psychological assessment at 12 weeks, 3 | baseline, 12 weeks
  • Mindfulness Attention Awareness Scale: A 15-item measure assessing mindfulness of moment to moment experience
Changes from baseline psychological assessment at 12 weeks, 4 | baseline, 12 weeks
  • Patient Health Questionnaire-9: A self-administered tool for assessing depression
Changes from baseline psychological assessment at 12 weeks, 5 | baseline, 12 weeks
  • Optimism. Revised Life Orientation Test: A questionnaire to assess individual's optimism and related to healthy aging seniors
Changes from baseline overall health surveys / physical frailty test at 12 weeks, 2 | baseline, 12 weeks
  • Barthel Index of Activities of Daily Living: A 10-item questionnaire for activities of daily living
Changes from baseline overall health surveys / physical frailty test at 12 weeks, 3 | baseline, 12 weeks
  • Pittsburgh Sleep Quality Index: A self-reported questionnaire that assesses sleep quality and disturbances
Changes from baseline overall health surveys / physical frailty test at 12 weeks, 4 | baseline, 12 weeks
  • Sarcopenia Questionnaire: This questionnaire will ask participants basic physical capability
Changes from baseline overall health surveys / physical frailty test at 12 weeks, 5 | baseline, 12 weeks
  • Mini Nutritional Assessment - Short Form: Assesses malnutrition, weight loss, and a lack of appetite
Knee Flexion and Extension Visual-Motor Reaction Time | baseline, after 12 weeks
  Subjects will be asked to kick up (quadriceps - knee extensors) or pull back (hamstrings - knee flexors) as soon as an arrow is displaced up or down, respectively.
Changes from baseline ultrasound-based bilateral anterior thigh muscle stiffness measurements at 12 weeks | baseline, 12 weeks
  Ultrasound probe will be placed at the mid-thigh (the quadriceps) during rest and knee extension strength force steadiness testing.

CONTACTS AND LOCATIONS:
Overall Officials: Takashi Nagai, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials